CLINICAL TRIAL: NCT00633997
Title: An Open-label, Multiple Dose Study to Assess the Steady-state Skin Concentrations and Pharmacokinetics of Vildagliptin 50 mg BID for 10 Days in Healthy Subjects and Patients With Type 2 Diabetes
Brief Title: Assessment of the Skin-concentration of Vildagliptin 50 mg Every 12 Hours for 10 Days in Healthy Subjects and Patients With Type 2 Diabetes
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: After analysis of the existing data, it was determined that additional skin biopsy samples would not be required to determine study outcome.
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CLAF237A2224
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2016-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes mellitus; type 2 diabetes; vildagliptin; pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Vildagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Healthy volunteers
  Interventions: Drug: Vildagliptin
- 2 (Experimental): Type II diabetics
  Interventions: Drug: Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin — 50 mg orally twice daily for 10 days (last dose morning of day 10)
  Other Names: LAF237 Galvus
  Arms: 1
Drug: Vildagliptin
  Arms: 2

SUMMARY:
This study will look at the skin accumulation of vildagliptin and its two major metabolites, LAY151 and LAF237-O-Glucuronide, after vildagliptin 50 mg given orally twice a day for 10 days in both healthy volunteers and patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers and patients with type 2 diabetes
* Non-smoking, Caucasian and African American, male and female (postmenopausal, surgically sterile or using double-barrier method of contraception) subjects between 30 and 65 years of age (inclusive)
* Type 2 diabetics on metformin and/or sufonylurea

Exclusion Criteria:

* History of type 1 diabetes or insulin use
* History of coagulation abnormalities
* History of abnormal heart conditions
* Pregnancy or breastfeeding

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Skin concentration of vildagliptin and its two metabolites, LAY151 and LAF237-O-Glucuronide, compared to the plasma concentration on Day 10 | Baseline (Day -1) to End of Study (Day 17 +/- 2 days)

SECONDARY OUTCOMES:
10 day's treatment with vildagliptin 50 mg orally twice daily on hematology, blood chemistry and physical exams in healthy volunteers and patients with type 2 diabetes | Baseline (Day -1) to End of study (Day 17 +/- 2 days)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis investigator site
Locations (1):
- Novartis Investigator Site, Baltimore, Maryland, United States

REFERENCES:
- See also: Results for CLAF237A2224 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2802